CLINICAL TRIAL: NCT05802407
Title: The Value of Molecular Residual Disease Monitoring Based on ctDNA in Resected Pancreatic Cancer
Acronym: MAP-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K3378-02
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Cancer; Resectable Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD-guided (Experimental): Patients with elevated MRD from baseline at the first imaging assessment but without radiographic progressive disease will receive a later-line therapy.
  Interventions: Drug: Later-line therapy
- Routine treatment (No Intervention): Patients with elevated MRD from baseline at the first imaging assessment but without radiographic progressive disease will continued their current therapy.

INTERVENTIONS:
Drug: Later-line therapy — Another chemotherapy regimen, targeted therapy, or immunotherapy
  Arms: MRD-guided

SUMMARY:
The goal of this clinical trial is to explore the value of molecular residual disease (MRD) monitoring based on ctDNA in resected pancreatic cancer. The main questions it aims to answer are:

* prognostic value of baseline MRD;
* the role of MRD dynamic changes after treatment in guiding treatment. Peripheral blood derived from participants will be obtained for MRD test before adjuvant chemotherapy initiation and at the first imaging assessment after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with pancreatic cancer who had undergone curative-intent surgery (R0 or R1 resection);
* both sexes, age ≥18 years old;
* ECOG performance status score ≤2;
* the expected survival time was ≥3 months.

Exclusion Criteria:

* a known diagnosis of pancreatic cancer other than ductal adenocarcinoma;
* treated with any systemic antitumor treatment before first-line chemotherapy onset;
* died or lost to follow-up within one month after the initiation of adjuvant chemotherpay;
* combined with other primary malignances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Baseline until death from any cause (up to approximately 36 months)
  The date of adjuvant chemotherpay initiation to tumor recurrence, local-regional or distant metastases, or death due to any cause.

SECONDARY OUTCOMES:
Overall survival | Baseline until death from any cause (up to approximately 60 months)
  The date of adjuvant chemotherpay initiation to death due to any cause.

OTHER OUTCOMES:
The prognostic value of MRD | Baseline until death from any cause (up to approximately 60 months)
  The prognostic value of baseline MRD and dynamic MRD changes
The prognostic role of targeted therapy selected based on MRD | Baseline until death from any cause (up to approximately 60 months)
  The prognostic role of targeted therapy selected based on MRD

CONTACTS AND LOCATIONS:
Overall Officials: Chunmei Bai, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Medical Oncology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided